CLINICAL TRIAL: NCT05260528
Title: An ALFA 2101 Multicenter Randomized Phase II Study: CPX-351 Versus Intensive Chemotherapy in Patients With de Novo Intermediate or Adverse Risk AML Stratified by Genomics
Brief Title: CPX-351 vs Intensive Chemotherapy in Patients With de Novo Intermediate or Adverse Risk AML Stratified by Genomics
Acronym: ALFA2101
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-PP-26
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: CPX-351; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Active Comparator)
  Interventions: Drug: Cytarabine and Idarubicin
- Investigational arm (Experimental)
  Interventions: Drug: CPX-315

INTERVENTIONS:
Drug: Cytarabine and Idarubicin — Induction 1: Cytarabine 200 mg/m2 i.v. (continuously) d1-7 + Idarubicin 12mg/m2 d1, 2, 3 i.v (60 min)
  Induction 2: Cytarabine 1500 mg/m2 i.v. q12h d1-3
  Consolidation: Cytarabine 1500 mg/m2 i.v. q12h d1-3
  Arms: Standard arm
Drug: CPX-315 — Induction 1:CPX-351 44 mg/m2 daunorubicin / 100 mg/m2 cytarabine i.v. (90 min) d1,3,5
  Induction 2: CPX-351 44 mg/m2 daunorubicin / 100 mg/m2 cytarabine i.v. (90 min) d1,3
  Consolidation therapy:CPX-351 29 mg/m2 daunorubicin / 65 mg/m2 cytarabine i.v. (90 min) d1,3
  Arms: Investigational arm

SUMMARY:
The trial is a randomized, open-label phase II study comparing CPX-351 vs conventional intensivechemotherapy in patients with newly diagnosed de novo AML and intermediate- or adverse-risk genetics (according to 2017 ELN criteria)

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous hematologic malignancy characterized by clonal expansion of myeloid blasts.

Interestingly comparing de novo and stringently defined secondary AMLs occurring after a documented phase of MDS, Lindsley et al. could identify among de novo AMLs a molecular subgroup, termed 'secondary-type AML', defined by mutations in either SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR and/or STAG2 genes. Among de novo AML patients, 33.3% had secondary-type mutations.

It has been shown that patients older than 60 years of age harboring secondary-type AML, as defined by this 8-gene molecular signature, had inferior outcome to those without 'secondary-type' mutations when treated with conventional 7+3 chemotherapy, combining cytarabine and an anthracycline (ALFA 1200 study). This was notably true among patients with 'intermediate-risk' disease per European LeukemiaNet criteria.

The incidence of 'secondary-type' AML mutations increases with age and with cytogenetic risk category. Notably, roughly 50% of de novo AML patients with intermediate risk older than 50 years of age harbor such secondary-type mutations, New therapeutic options are thus necessary in patients older than 50 years with de novo AML classified adverse risk but also intermediate risk and associated to secondary-type mutation

This study will evaluate the rate of MRD negative remissions with CPX-351 used as induction and consolidation therapy according to its marketing authorization (AMM), as compared to intensive chemotherapy in a population of non-MRC AMLs enriched in secondary-like mutations. In addition,P-gp activity will be explore as a putative biomarker.

Duration of the enrollment period: 36 months Duration of treatment: 6 months Duration of the participation for a patient: 18 months (post randomization) (including approximately 6 months treatment, and 12 months of post-treatment follow up) Overall duration of the study: 58 months including the analysis of the results

ELIGIBILITY:
Inclusion Criteria:

1. De novo AML
2. No MRC-defining cytogenetic lesion
3. No t(15;17), t(8;21), inv(16) or t(16;16)
4. No NPM1 gene mutation
5. No FLT3 mutated AML (FLT3 ITD or TKD)
6. Not previously treated except for short course hydroxyurea in patients presenting with high WBC count and/or tumor symptoms,
7. Age ≥ 50 years,
8. Performance status ≤ 2 (ECOG grading),
9. Patient must have adequate organ function as indicated detailed with laboratory values in the section IV of the protocol
10. Female patient of childbearing potential with a negative serum pregnancy test (β-hCG) within 72 hours prior to receiving the first dose of CPX-351 or 7+3. Female patient who is not actively breastfeeding at the time of study entry.
11. Female patient is either post-menopausal, free from menses for > 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy, or agrees to not become pregnant throughout the study, starting with study screening
12. Male patient agrees to use an adequate method of contraception for the duration of the study. Men should be advised not to father a child while receiving CPX-351 or 7+3 and for 3 months after the last dose of study treatment .
13. Patient is available for periodic blood sampling, study related assessments, and appropriate clinical management at the treating institution for the duration of the study.
14. Patient has the ability to understand and willingness to sign an informed consent form indicating the investigational nature of the study.
15. Patient registered to the French Social Security.

Exclusion Criteria:

1. Prior history of documented MDS, MPN or MDS/MPN, tAML
2. Prior history of radiation therapy or chemotherapy for a solid tumor or lymphoma (exceptions to be considered: local radiotherapy for prostate cancer)
3. Patient has active and uncontrolled infection.
4. Patient has uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including but not limited to the following: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pancreatitis, or psychiatric or social conditions that may interfere with patient compliance.
5. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug.
6. Patient has known human immunodeficiency virus (HIV) infection or HIV-related malignancy.
7. Patient has clinically active hepatitis B or hepatitis C infection.
8. Patient has a known allergy or hypersensitivity to any component of CPX-351, idarubicin or cytarabine.
9. Patient with a "currently active" second malignancy, other than nonmelanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >1 year or are considered by their physician to be at less than 30% risk of relapse.
10. Patients with clinical evidence of CNS leukemia.
11. Cardiac ejection fraction <50% or considered as abnormal by echocardiography or multi-gated acquisition (MUGA) scan.
12. Patient is pregnant or breastfeeding within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in the proportion of patients achieving deep remission (CR)/(CRi) with a standardized flow based MRD in the BM aspirate using the LAIP/Dfn method after the 1st induction | 28-56 days

SECONDARY OUTCOMES:
Rate of CR/CRi with a flow based MRD in the BM aspirate using the LAIP/Dfn method | 28-56 days
Analysis of rate of flow-based MRD quantified in the bone marrow according to both the LAIP/DfN method and the LSC method | 10-13 weeks
Analysis of flow-based MRD quantified according to both LAIP/DfN method and the LSC methods | 10-13 weeks
Overall response rate, and CR and CRi rates | 28-56 days
Cumulative incidence of allogeneic HSCT | 4.5 years
Early mortality at D30, D60, D100 | day 100
Overall Survival (with and without censoring at allogeneic HSCT) | 4.5 years
Relapse-Free Survival (with and without censoring at allo-HSCT) | 4.5 years
Event-Free Survival (with and without censoring at allo-HSCT) | 4.5 years
Cumulative Incidence of Relapse (with and without censoring at allo-HSCT) | 4.5 years
Analysis of Hematological and non-hematological toxicity profile and safety using the NCI- common toxicity criteria (CTCAE) version 5.0 of November 2017 | 4.5 years
Analysis of duration of hospitalization during induction and consolidation cycles | 6 months
Analysis of changes of the genomic landscape with the treatment | 6 months
Analysis of the somatic mutations (documented with their allele frequency) associated with AML and OS, RFS | 4.5 years
QoL EORTC QLQ-C30 ( core quality of life questionnaire developped by European Organization for Research and treatment of Cancer), Self assessment by patients | 6 months
  The EORTC QLQ-C30nsubscales scores are tranformed to a 0 to 100 scale, with higher score on functionnal scales indicating better function and higher scores on sumptom scales indicating worse symptoms
Analysis of secondary-type mutational profile at screening as determined by Lindsley et al | 6 months
  Exploratory objectives
Analysis of entralized functional flow cytometry assays at baseline carried on peripheral blood or bone marrow aspirate | 6 months
  Exploratory objectives
Analysis of Flow MRD | 6 months
  Exploratory objectives

CONTACTS AND LOCATIONS:
Locations (30):
- France (30):
  - CHU Amiens Picardie site Sud, Amiens
  - CH Avignon, Avignon
  - CHRU Jean Minjoz, Besançon
  - Centre Hospitalier de Béziers, Béziers
  - Hôpital Avicenne APHP, Bobigny
  - Institut d'hématologie de Basse Normandie (IHBN), Caen
  - Hôpital d'Instruction des Armée (HIA), Clamart
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien (CHSF), Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier de Versailles, Site André Mignot, Le Chesnay
  - Hôpital Claude HURIEZ, CHU Lille, Lille
  - CHU de Limoges, Limoges
  - Hoptial de la Conception APHM, Marseille
  - CHR Metz-Thionville Site Mercy, Metz
  - Groupe hospitalier de la région de Mulhouse et Sud-Alsace, Hôpital Emile Muller, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - Institut de cancérologie du Gard, Nîmes
  - CHR Orléans, Orléans
  - Hopital Necker, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Saint-Louis, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Hopital Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif